CLINICAL TRIAL: NCT01971489
Title: A Phase I Study of the PI3-Kinase Inhibitor BKM120 in Combination With Gemcitabine and Cisplatin in Patients With Advanced Solid Tumors
Brief Title: Buparlisib, Gemcitabine Hydrochloride, and Cisplatin in Treating Patients With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 240413; NCI-2013-01941 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 240413 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Adult Solid Neoplasm; Recurrent Non-Small Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — NVP-BKM120; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (buparlisib, gemcitabine hydrochloride, cisplatin) (Experimental): Patients receive buparlisib PO QD on days 1-21, gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, and cisplatin IV over 2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Buparlisib; Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Buparlisib — Given PO
  Other Names: BKM120; PI3K Inhibitor BKM120
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial studies the side effects and the best doses of buparlisib, gemcitabine hydrochloride, and cisplatin in treating patients with solid tumors that have spread to other places in the body. Buparlisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine hydrochloride and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving buparlisib, gemcitabine hydrochloride, and cisplatin may be a better treatment for solid tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the dose-limiting toxicities, maximally tolerated dose, and identify the recommended Phase II dose (RP2D) of the combination of BKM120 (buparlisib), gemcitabine (gemcitabine hydrochloride), and cisplatin in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. To describe safety and tolerability of the combination of BKM120, gemcitabine, and cisplatin in patients with advanced solid tumors.

II. To describe preliminary evidence of efficacy with this combination. III. To describe any pharmacokinetic (PK) effect of gemcitabine and cisplatin on the plasma concentrations of BKM120.

IV. To evaluate phosphatidylinositol-4, 5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) mutations as predictive biomarkers of efficacy for the combination.

V. To evaluate PIK3CA polymorphisms and polymorphisms in BKM120 transport and metabolism as predictors of toxicity and/or efficacy.

OUTLINE: This is a dose-escalation study.

Patients receive buparlisib orally (PO) once daily (QD) on days 1-21, gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1 and 8, and cisplatin IV over 2 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of solid malignancy
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Life expectancy of >= 12 weeks
* Platelet count >= 150 x 10^9/L
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Hemoglobin (Hgb) >= 9 g/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 1.5 upper limit normal (ULN), or < 3 x ULN if liver metastases are present
* Serum total bilirubin =< ULN or 1.5 x ULN if liver metastases are present or total 3 x ULN with direct bilirubin =< ULN in patients with well documented Gilbert syndrome
* Calculated or measured creatinine clearance >= 60 mL/min
* Fasting plasma glucose < 120 mg/dL
* Magnesium >= the lower limit of normal
* Lipase =< 1.5 ULN
* Women of childbearing potential must have a negative pregnancy test performed within 7 days prior to the start of study drug
* Male and female subjects of child-bearing potential must agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during the study and for 90 days after last investigational drug dose received
* Subject or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* For dose expansion cohort, patients must have histologic or cytologic confirmed non-small cell lung cancer that are not curable

Exclusion Criteria:

* Previous anti-cancer chemotherapy, immunotherapy or investigational agents < 4 weeks, or palliative radiation < 2 weeks prior to the first day of study treatment, or who have not recovered to grade 1 or better from related side effects of such therapy (except alopecia); patients who receive gamma knife radiosurgery for brain metastases are eligible if procedure was performed > 2 weeks before treatment is started, is clinically stable and has been on stable low dose corticosteroid treatment (e.g., dexamethasone 2 mg/day, prednisolone 12 mg/day for at least 14 days before start of study treatment are eligible); ongoing hormonal therapies (luteinizing hormone-releasing hormone [LHRH] antagonists, megestrol) are allowed
* Previous treatment with a phosphatidylinositol 3-kinase (P1-3K) inhibitor
* Patients who have taken herbal medications and certain fruits within 7 days prior to starting study drug; herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng; fruits include the cytochrome P450, family 3, subfamily A (CYP3A) inhibitors Seville oranges, grapefruit, pummelos, or exotic citrus fruits
* Patient has a known hypersensitivity to any of the excipients of BKM120
* Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects
* Patient is currently receiving increasing or chronic treatment (> 5 days) with corticosteroids or another immunosuppressive agent, as chronic administration of corticosteroids (> 5 days) can induce cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4)

  * The following uses of corticosteroids are permitted: single doses; e.g. with standard premedication for taxanes; topical applications (e.g., rash), inhaled sprays (e.g., obstructive airways diseases), eye drops or local injections (e.g., intra-articular)
* Patient is being treated at start of study treatment with any of the following drugs:

  * Drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A4 including herbal medications
  * Drugs with a known risk to induce Torsades de Pointes
  * Note: The patient must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the treatment is initiated; switching to a different medication prior to starting study treatment is allowed
* Patient is currently receiving warfarin or other Coumarin derived anti-coagulant, for treatment, prophylaxis or otherwise; therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed
* Patients who have other concurrent severe and/or uncontrolled medical conditions that would, in the investigator's judgment, contraindicate patient participation in the clinical study (eg. active or uncontrolled severe infection, chronic active hepatitis, immunocompromised, acute or chronic pancreatitis, uncontrolled high blood pressure, interstitial lung disease, etc.)
* Patient has a known history of human immunodeficiency virus (HIV) infection (testing not mandatory) infection
* Patient has any of the following cardiac abnormalities:

  * Symptomatic congestive heart failure

    * History of documented congestive heart failure (New York Heart Association functional classification III-IV), documented cardiomyopathy
    * Left ventricular ejection fraction (LVEF) < 50% as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO)
  * Myocardial infarction =< 6 months prior to enrollment
  * Unstable angina pectoris
  * Serious uncontrolled cardiac arrhythmia
  * Symptomatic pericarditis
  * Corrected QT interval using Fridericia's formula (QTcF) > 480 msec on the screening electrocardiogram (ECG) (using the QTcF formula)
  * Currently receiving treatment with medication that has a known risk to prolong the QT interval or inducing Torsades de Pointes, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Patient has a score >= 12 on the Patient Health Questionnaire (PHQ)-9 questionnaire
* Patient selects a response of "1, 2 or 3" to question number 9 on the PHQ-9 questionnaire regarding potential for suicidal thoughts or ideation (independent of the total score of the PHQ-9)
* Patient has a General Anxiety Disorder (GAD)-7 mood scale score >= 15
* Patient has a medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others), or patients with active severe personality disorders (defined according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition [DSM-IV]) are not eligible; Note: for patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous 6 weeks prior to start of study drug
* Patient has >= Common Terminology Criteria for Adverse Events (CTCAE) grade 3 anxiety
* Patient has other prior or concurrent malignancy (except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, early gastric or GI cancer resected completely by endoscopy procedures or any other cancer from which the patient has been disease free for >= 3 years)
* Patient has a history of non-compliance to medical regimen or inability to grant consent
* Patient is concurrently using other approved or investigational antineoplastic agent
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (> 5 mIU/mL); patients with elevated hCG at baseline that is judged to be related to the tumor are eligible if hCG levels do not show the expected doubling when repeated 5-7 days later, or pregnancy has been ruled out by vaginal ultrasound
* Patient who does not apply highly effective contraception during the study and through the duration as defined below after the final dose of study treatment:

  * Sexually active males should use a condom during intercourse while taking drug and for 8 weeks after the final dose of study treatment and should not father a child in this period, but may be recommended to seek advice on conservation of sperm; a condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid
  * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study and through at least 4 weeks after the final dose of study treatment
  * Highly effective contraception is defined as either:

    * Total abstinence: when this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception)
    * Female sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate); (for female study subjects, the vasectomized male partner should be the sole partner for that patient)
    * Use a combination of the following:

      * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
      * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
      * Note: hormonal contraception methods (e.g. oral, injected, and implanted) are not allowed
* Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago; for women with therapy-induced amenorrhea, oophorectomy or serial measurements of follicle-stimulating hormone (FSH) and/or estradiol are needed to ensure postmenopausal status; NOTE: ovarian radiation or treatment with a luteinizing hormone-releasing hormone (LH-RH) agonist (goserelin acetate or leuprolide acetate) is not permitted for induction of ovarian suppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) using the National Cancer Institute (NCI) CTCAE version 4.0 | Up to 21 days
  Adverse events will be coded and evaluated for severity using NCI-CTCAE, version 4.0 and will be summarized by system organ class and preferred term.
Maximum-tolerated dose (MTD) defined as the maximum dose level at which less than or equal to 1 out of 6 patients have DLTs using NCI CTCAE version 4.0 | Up to 21 days

SECONDARY OUTCOMES:
Disease control rate using RECIST (CR, PR, and SD) | Up to 30 days after completion of study treatment
Objective response rate (ORR) calculated as the number of patients with a confirmed complete response (CR) or partial response (PR) divided by the total number of patients using Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 30 days after completion of study treatment
  Tumor response will be summarized for the evaluable patient population, and the 95% confidence interval for ORR (CR+PR) will be presented.
PIK3CA mutations | Up to 30 days after completion of study treatment
  Will be assessed as potential predictive biomarkers of efficacy for the combination.
PIK3CA polymorphisms | Up to 30 days after completion of study treatment
PK effect of gemcitabine hydrochloride and cisplatin on buparlisib | Pre-dose and at 0.5, 1, 2, and 4 hours post-dose on day 21 of course 1, and pre-dose and 0.5, 1, 2, and 4 hours post-dose on day 1 of course 2 (or day 3 of course 2 for the 2 days off, 5 days on dosing schedule)
  PK parameters include time to reach maximum concentration (Tmax), maximum concentration (Cmax), clearance (CL), half-life (T1/2), area under the curve (AUC)0-infinity, and AUC0-t for the dosing interval following multiple dose administration.
Polymorphisms in buparlisib transport and metabolism | Up to 30 days after completion of study treatment
  Will be assessed as potential predictors of toxicity and/or efficacy.
RECIST response | Up to 30 days after completion of study treatment
  The number and percent of patients qualifying for each RECIST response category (CR, PR, stable disease [SD], and progressive disease [PD]).

CONTACTS AND LOCATIONS:
Overall Officials: Alex Adjei, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States